CLINICAL TRIAL: NCT07059130
Title: Evaluating the Efficacy and Safety of Mirikizumab in Adults Over 60 With Moderate to Severe Crohn's Disease and Ulcerative Colitis: A Phase IV Multicenter Interventional Study
Brief Title: Evaluating the Efficacy and Safety of Mirikizumab in Adults Over 60 With Moderate to Severe Crohn's Disease and Ulcerative Colitis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rubix LS (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REX201233
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Crohn Disease (CD); Crohns Disease; Ulcerative Colitis (UC)
Keywords: Mirikizumab; Crohn's Disease; Ulcerative Colitis; Clinical remission; Elderly; Biomarkers; IBD
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — mirikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mirikizumab Treatment Group (Experimental): Participants aged 60 years and older with moderate-to-severe Crohn's Disease (CD) or Ulcerative Colitis (UC) will receive Mirikizumab administered according to FDA-approved dosing guidelines. All enrolled participants will be assigned to this single intervention group for the entire study duration.
  Interventions: Biological: Mirikizumab

INTERVENTIONS:
Biological: Mirikizumab — Mirikizumab will be administered to participants according to FDA-approved dosing guidelines for moderate-to-severe Crohn's Disease and Ulcerative Colitis. Participants will receive scheduled doses throughout the study period at predefined intervals. Clinical assessments, patient-reported outcomes, biomarker analyses, and safety monitoring will occur at baseline and at Weeks 12, 24, and 48.
  Other Names: Mirikizumab Treatment Group

SUMMARY:
This research study looks at how safe and effective a medicine called Mirikizumab is for treating older adults (aged 60 and above) who have moderate to severe Crohn's disease (CD) or ulcerative colitis (UC). These two conditions, known as inflammatory bowel diseases (IBD), cause inflammation (swelling and irritation) in the digestive tract. Older adults with these conditions often have other health issues and face increased risks and complications, making it challenging for them to use certain treatments.

Mirikizumab is already approved by the FDA for adults with IBD, but there's limited information about how well it works specifically for older adults. This study aims to fill that gap by seeing if Mirikizumab can help these patients safely manage their condition.

The study plans to enroll around 150 people from various locations across the United States. Everyone participating will receive Mirikizumab according to the standard, FDA-approved guidelines.

The main goal is to see how many participants achieve clinical remission, meaning their symptoms significantly improve or disappear, after 24 weeks of treatment. Researchers will also look at whether this remission lasts up to 48 weeks, how well symptoms are controlled without steroids, how treatment affects indicators of inflammation (such as blood tests), and how the participants feel overall based on their own reports.

The safety of Mirikizumab will also be closely monitored throughout the study by regularly checking for any side effects.

This study hopes to provide clearer information to help older adults with IBD and their doctors make better treatment decisions, ultimately improving health outcomes and quality of life.

DETAILED DESCRIPTION:
This study is a Phase IV clinical trial designed specifically to examine how older adults (aged 60 years and above) respond to Mirikizumab, a biologic treatment approved by the FDA for inflammatory bowel disease (IBD). Recognizing the limited clinical trial representation of older patients, this study aims to provide essential evidence on treatment effectiveness, safety, and patient experience within this specific age group, addressing an existing knowledge gap in clinical practice.

The trial will enroll approximately 150 adult participants diagnosed with moderate-to-severe Crohn's Disease (CD) or Ulcerative Colitis (UC) across multiple academic and community healthcare settings within the United States. Enrolled participants will undergo treatment with Mirikizumab administered strictly in accordance with FDA-approved dosing guidelines, without comparator or placebo groups.

Key measures of clinical improvement include standardized, validated scoring systems: the Crohn's Disease Activity Index (CDAI) for CD participants and the Mayo Score for UC participants. Additionally, validated biomarkers indicative of disease activity (e.g., CRP, fecal calprotectin) and standardized patient-reported outcome measures (Inflammatory Bowel Disease Questionnaire [IBDQ]) will be evaluated at specified intervals.

Participants will attend scheduled visits at baseline (Week 0), and subsequently at Weeks 12, 24, and 48. At each visit, researchers will assess clinical status, collect biological samples for biomarker analysis, review patient-reported outcomes, and systematically document any side effects or adverse events associated with treatment.

Safety will be carefully monitored by an independent Data Monitoring Committee (DMC), which will review collected safety data semi-annually. Procedures for adverse event reporting are rigorous, following strict regulatory guidelines to ensure participant safety.

Comprehensive strategies to retain and support study participants include regular follow-up contacts, adherence monitoring, patient education initiatives, and flexible scheduling for convenience.

Data collected throughout the trial will be securely managed using electronic data capture systems with strict confidentiality and quality control protocols in place. Statistical analyses will involve standard intention-to-treat (ITT) methods and mixed-model statistical approaches to accurately determine treatment effectiveness and safety outcomes.

Ultimately, the findings from this trial aim to inform clinical care guidelines for older adults with IBD and enhance clinical decision-making by providing robust, real-world evidence specific to the aging population.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 60 years or older at the time of enrollment.

Diagnosed with moderate-to-severe Crohn's Disease (CDAI score ≥220) or moderate-to-severe Ulcerative Colitis (Mayo Score ≥6).

Capable of providing informed consent for participation in the study.

Exclusion Criteria:

History of recent major gastrointestinal surgery within 3 months prior to enrollment.

Active infection requiring antibiotic or antiviral treatment at the time of enrollment.

Active malignancy or a history of malignancy within the past 5 years. (Exception: Participants with fully resected basal cell carcinoma or squamous cell carcinoma of the skin, with no metastatic disease for at least 3 years, are eligible.)

Current use or recent participation (within 30 days) in another clinical trial involving investigational therapies.

Contraindication or known hypersensitivity to biologic medications, specifically Mirikizumab.

Active cardiovascular disease, including:

Unstable angina, myocardial infarction, or cardiovascular procedures within the past 6 months.

Uncontrolled hypertension (systolic ≥160 mmHg or diastolic ≥100 mmHg despite treatment).

Congestive heart failure (NYHA Class III or IV).

Clinically significant arrhythmias or other unstable cardiovascular conditions.

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-16 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Clinical Remission at Week 24 | 24 weeks
  Clinical remission is defined as achieving either:
  Crohn's Disease Activity Index (CDAI) score less than 150 (for participants with Crohn's Disease), or
  Mayo Score of 2 or less (for participants with Ulcerative Colitis).

CONTACTS AND LOCATIONS:
Locations (1):
- Rubix LS, Lawrence, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) sharing is currently undecided. Any future requests for data sharing will be carefully considered and reviewed by the sponsor (Rubix LS) on a case-by-case basis, taking into account the nature of the request, ethical considerations, privacy of study participants, and potential scientific value of data sharing.